CLINICAL TRIAL: NCT02747615
Title: Efficacy of Preoperative Autologous Blood Donation and Tranexamic Acid in Revision Total Hip Arthroplasty: a Randomized Controlled Trial
Brief Title: Efficacy of Preoperative Autologous Blood Donation and Tranexamic Acid in Revision Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, MD, Lecturer of Anesthesia and Intensive Care Medicine, Ain Shams University Hospitals, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 586
Record Dates: First submitted 2016-04-03; First posted 2016-04-22 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Revision Total Hip Arthroplasty (RTHA)
Keywords: Autologous blood donation, allogeneic blood transfusion

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Control group (n=30) (Other): The control group, which consisted of 30 patients who were transfused only allogeneic blood.
  Interventions: Other: transfused only allogeneic blood.
- Preoperative blood donation (n=30) (Active Comparator): the study group including 30patients who were transfused pre-operatively donated autologous blood, either during surgery or after it.
  Interventions: Other: transfused pre-operatively donated autologous blood.; Drug: intravenous tranexamic acid (TXA) infusion

INTERVENTIONS:
Other: transfused pre-operatively donated autologous blood. — Pre-operative autologous donation for minimising perioperative allogeneic blood transfusion
  Other Names: Pre-operative autologous donation
  Arms: Preoperative blood donation (n=30)
Drug: intravenous tranexamic acid (TXA) infusion — Intravenous tranexamic acid is a safe pharmacological treatment to reduce blood loss and transfusion requirements in patients undergoing major orthopedic surgery.
  Other Names: Kapron®
  Arms: Preoperative blood donation (n=30)
Other: transfused only allogeneic blood.
  Arms: Control group (n=30)

SUMMARY:
Sixty patients aged between 60 and 75 years old of both sex of ASA physical status I and II were included in this randomized study who were divided into the study group of 30 patients who had been transfused autologous blood and the control group of 30 patients who had been transfused only allogeneic blood. Parenteral iron preparation was given to all patients of the study group after each donation. Intraoperatively all patients of the study group received 2 grams of intravenous tranexamic acid. This study was conducted through the laboratory analysis of the hemoglobin and the hematocrit values during blood donation and for both groups in the pre-operative and the post-operative period and the assessment of the amount of transfused blood units in both groups.

DETAILED DESCRIPTION:
A total of 60 patients were included in this randomized study that were divided into a study group of 30 patients, who had been transfused autologous blood and a control group of 30 patients who had been transfused only allogeneic blood. Parenteral iron preparation was given to all patients of the study group after each donation. Intraoperatively all patients of the study group received 2 g of intravenous TXA.

This study was conducted through laboratory analysis of hemoglobin and hematocrit values during blood donation and for both groups in the preoperative and the postoperative period and the assessment of the amount of transfused blood units in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Elective revision total hip replacement surgery was performed in 60 patients aged between 60 and 75 years old of both sex of ASA physical status I and II of 70-90 kg body weight and height 160-180 cm.

Exclusion Criteria:

* This study excluded cases of revision total hip arthroplasty (RTHA) for infection or fractures as well as early revisions for dislocations secondary to implant malposition. Preoperative autologous blood donation was not done in patients with cardiac decompensation, severe hemodynamic problems, respiratory insufficiency, severe defect of central nervous system, active infection, blood disease or coagulopathies.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group (n=30): The control group, which consisted of 30 patients who were transfused only allogeneic blood.
  transfused only allogeneic blood.
- Preoperative Blood Donation (n=30): the study group including 30patients who were transfused pre-operatively donated autologous blood, either during surgery or after it.
  transfused pre-operatively donated autologous blood.
  intravenous tranexamic acid (TXA) infusion
Period: Overall Study
Arm/Group | Control Group (n=30) | Preoperative Blood Donation (n=30)
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group (n=30) | Preoperative Blood Donation (n=30) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (4.4) | 67.4 (4.1) | 67.6 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 11 | 14 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Transfused Allogeneic Blood Units (in Digits).
Time Frame: 48-72 hours after surgery.
Measure: Median (Inter-Quartile Range); unit: units
Arm/Group | Control Group (n=30) | Preoperative Blood Donation (n=30)
Number analyzed (Participants) | 30 | 30
units | 2.0 [1.0 to 3.0] | 0.0 [0.0 to 1.0]

2. Secondary Outcome: Our Secondary Outcome Measure Was to Assess the Post-operative Hospital Stay (Days).
Time Frame: 48-72 hours after surgery.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control Group (n=30) | Preoperative Blood Donation (n=30)
Number analyzed (Participants) | 30 | 30
days | 5.27 (1.11) | 3.20 (0.41)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 24 hours postoperatively.
Arm/Group | Control Group (n=30) | Preoperative Blood Donation (n=30)
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No